CLINICAL TRIAL: NCT01038401
Title: Characterization of the Residual Replication of HIV-1 in the Gut-associated Lymphoid Tissue in Patients Receiving Effective Highly Active Antiretroviral Therapy: the ANRS EP 44 Study
Brief Title: Residual Replication of HIV-1 in the Gut Associated Lymphoid Tissue (GALT) of Patients on Highly Active Antiretroviral Therapy (HAART): the ANRS EP 44 Study
Acronym: EP 44
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Lucie Marchand/Project manager, French National Agency for Research on AIDS and Viral Hepatitis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-A00239-46
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: HIV Infection
Keywords: HIV infection; HAART; Viral DNA test positive-10063306; Blood HIV RNA 10049826; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-1-infected patients on effective HAART (Other)
  Interventions: Procedure: GI endoscopy and GALT biopsies; Biological: A sample of venous blood will also be collected
- Non Infected HIV Volunteers (Other)
  Interventions: Procedure: GI endoscopy and GALT biopsies; Biological: A sample of venous blood will also be collected

INTERVENTIONS:
Procedure: GI endoscopy and GALT biopsies — This project aims to characterize the residual replication of HIV-1 in subjects on HAART, particularly in the gut-associated lymphoid tissue (GALT)
Biological: A sample of venous blood will also be collected — These samples of blood will be use to characterize the residual viral populations on effective HAART in three compartments, plasma, monocytes, and GALT

SUMMARY:
HIV-1 cannot be eradicated from infected individuals by current antiretroviral regimens. Cellular reservoirs and tissue sanctuary sites allow latent HIV-1 persistence and ongoing low-level virus replication. This project aims to characterize the residual replication of HIV-1 in subjects on antiretroviral therapy, particularly in the gut-associated lymphoid tissue.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) successfully controls HIV-1 replication in most individuals, resulting in substantial immune restoration and decreased morbidity and mortality. However HIV-1 cannot be eradicated from infected individuals by current regimens. Cellular reservoirs and tissue sanctuary sites allow latent HIV-1 persistence and ongoing low-level virus replication, despite maximum virus suppression on HAART. This project aims to characterize the residual replication of HIV-1 in subjects on HAART, particularly in the gut-associated lymphoid tissue (GALT). A group of 20 HIV-1-infected patients on effective HAART will undergo GI endoscopy and GALT biopsies will be taken. A sample of venous blood will also be collected. These samples will be use to characterize the residual viral populations on effective HAART in three compartments, plasma, monocytes, and GALT. HIV-1 coreceptor usage and its evolution on HAART will be characterized in virus reservoirs. This project could provide further insights into the residual replication of HIV-1 in subjects receiving HAART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection (ELISA and western-blot tests)
* Continuous antiretroviral therapy >= 12 months
* Plasma HIV-1 RNA =< 40 copies/ml >= 6 months
* Indication of gastro-intestinal endoscopy
* Age >= 18-year old
* Physical examination
* Informed consent

Exclusion Criteria:

* Plasma HIV-1 RNA > 40 copies/ml in the last 6 months
* Involvement in a HIV vaccine study
* Treatment with interferon-alpha or PEG- interferon-alpha in the last 6 months
* Treatment with interleukin-2 in the last 6 months
* Decompensated cirrhosis
* Abnormal hemostasis tests
* Inflammatory bowel disease ; coeliac disease
* Lymphoma
* Blood transfusion in the last 6 months
* Absence of social security (health insurance)
* Pregnant or breastfeeding woman
* Incapable adult

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Correlation between HIV-1 viral load and CD4+ T lymphopenia in the GALT.

SECONDARY OUTCOMES:
HIV-1 DNA load in the GALT vs blood CD4+ T cells
HIV-1 tropism in the GALT vs blood CD4+ T cells
Characterization of residual HIV-1 in the plasma < 40 copies/ml
Characterization of HIV-1 DNA in blood monocytes

CONTACTS AND LOCATIONS:
Overall Officials: MASSIP Patrice, Principal Investigator — University Hospital, Toulouse
Locations (1):
- ANRS center from Toulouse, Toulouse, France

REFERENCES:
- See also: Related Info — http://anrs.fr